CLINICAL TRIAL: NCT06761924
Title: Predictors of Response to Ultrasound-Guided Thoracic Paravertebral Nerve Block in Patients With Herpetic Neuralgia
Brief Title: Predicting Ultrasound-Guided Thoracic PVB Success in Herpetic Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMBSUREC/01092024/Yousef
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Patient Satisfaction
Keywords: Thoracic paravertebral nerve block; Herpetic neuralgia; Pain relief
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB group (Active Comparator): patients will receive ultrasound-guided TPVB with 25 mg bupivacaine 0.5%, plus 8 mg dexamethasone (10 mL volume)
  Interventions: Procedure: Ultrasound-Guided Thoracic Paravertebral nerve block
- Control group (Placebo Comparator): ultrasound-guided TPVB with 10 mL of saline without knowing which treatment they are receiving, maintaining blinding throughout the study
  Interventions: Procedure: Ultrasound-Guided Thoracic Paravertebral nerve block

INTERVENTIONS:
Procedure: Ultrasound-Guided Thoracic Paravertebral nerve block — The patients will receive ultrasound-guided TPVB with 25 mg bupivacaine 0.5%, plus 8 mg dexamethasone (10 mL volume)
  Arms: TPVB group
Procedure: Ultrasound-Guided Thoracic Paravertebral nerve block — ultrasound-guided TPVB with 10 mL of saline without knowing which treatment they are receiving, maintaining blinding throughout the study.
  Arms: Control group

SUMMARY:
This study aims to fill the knowledge gap by investigating the predictors of success for TPVB in patients with herpetic neuralgia. By identifying demographic, clinical, previous medications and procedural factors associated with positive outcomes, this research seeks to enhance the efficacy of TPVB and improve pain management strategies for patients suffering from herpetic neuralgia.

DETAILED DESCRIPTION:
Herpes zoster (HZ) is characterized by a unilateral dermatomal vesicular rash and severe discomfort along the affected dermatome. It is often caused by the reactivation of previously latent varicella zoster viruses (VZV) in cases of impaired cellular immunity.

According to recent population-based research , the overall incidence of HZ is almost 6.64/1000 person-years in the population aged 50 years or over, and it rises with age.

The most prevalent and severe side effect of HZ is post-herpetic neuralgia (PHN), which is commonly described as pain that lasts for 90 days after the rash first appears. Age-related increases in PHN incidence range from 5 to 30%, with patients over 50 having a higher risk if they have severe acute pain, a rash with many lesions, or strong prodromal symptoms.

Regretfully, there hasn't been a treatment that consistently reduces PHN discomfort up until now. Data from much research showed that patients may have significant clinical and financial burdens as a result of HZ and its consequences.

Analgesics are typically also needed, even though the availability of antiviral medications can speed up the end of viral shedding and quicken the healing of rash. Furthermore, it has no discernible effect on the development of PHN. As a result, it is crucial to start a methodical treatment plan that might have a preventative impact on PHN. It has been demonstrated that paravertebral nerve block is effective in treating acute pain in HZ patients, and it appears to have a greater antiviral treatment-induced reduction in PHN incidence.

Thoracic paravertebral block ( TPVB) involves the injection of local anesthetics and steroids adjacent to the thoracic vertebrae, resulting in the blockade of spinal nerves. This technique can provide segmental anesthesia and prolonged pain relief, making it a valuable tool in the anesthesiologist's repertoire. While TPVB is commonly used for postoperative analgesia in thoracic surgery, its application in managing herpetic neuralgia pain is relatively underexplored as the most recent evidence was published in 2023. Despite the potential benefits of TPVB in treating herpetic neuralgia, there is limited understanding of the factors that predict its success. Identifying these predictors could optimize patient selection and improve outcomes, but current literature on this topic is sparse.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from18 to 70 years
* Diagnosed with herpetic neuralgia.
* Able and willing to provide informed consent.
* ASA I - II
* One dermatomal affection
* Thoracic distribution

Exclusion Criteria:

* Contraindications to TPVB as ( Infection at site of injection, empyema , coagulopathy and neoplastic lesion occupying the paravertebral space)
* Known allergies to study medications (bupivacaine, Dexamethasone).
* Severe comorbidities that could interfere with study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale (NRS) | baseline , 24 hours , 2 weeks ,6 weeks , 3 months and 6 months post- intervention
  The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours. The average of the 3 ratings was used to represent the patient's level of pain over the previous 24 hours

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours,2 weeks ,6 weeks, 3 months and 6 months post- intervention.
  At baseline , 24 hours ,2week, 6week, 3 months and 6 months post- intervention using TreatmentSatisfaction Questionnaire for Medication (TSQM v1.4)

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt